CLINICAL TRIAL: NCT07008989
Title: Use of a Digital Memory Prosthetic to Support Autobiographical Memory in Down Syndrome
Brief Title: A VIRTUAL Three-month Intervention Study of the Effects of a Smartphone Application (HippoCamera) on Memory in Teens and Young Adults With Down Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston College (Other)
Collaborators: Massachusetts General Hospital (Other); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1R21HD114263 (NIH)
Record Dates: First submitted 2025-05-27; First posted 2025-06-06 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Memory Replay; HippoCamera
Keywords: Down syndrome; memory; hippocampus; technology
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: Following a baseline screening and memory test, participants will be randomly assigned to one group. During the first 12 weeks, one group will be assigned to the HippoCamera intervention and the other will serve as a control, receiving no intervention. After the first 12 weeks, the second group will receive the HippoCamera intervention.
  Within the HippoCamera application, half of all recorded events will be categorized as "baseline" memories, and half will be categorized as "replay" memories. Baseline memories are recorded, but never viewed by the participant again until the test at the end of the 12-week intervention. Replay memories are recorded, and then placed into a memory gallery. HippoCamera uses a research-based algorithm to select 5 memories from this gallery for participants to replay each day. Prior research has shown that this replay is associated with significant memory enhancements for replayed v. baseline memories for HippoCamera users from other populations.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate intervention (Experimental): During the first 12 weeks following enrollment, the Immediate Intervention group will engage in daily practice with the HippoCamera app. HippoCamera is a smartphone application that allows participants to record and replay important events in their daily lives. Based on principles from psychology and neuroscience, engaging in this daily practice may increase focus on memory-orientated practices in participants.
  Interventions: Behavioral: Memory replay
- Delayed Intervention (Other): During the first 12 weeks following enrollment, the Delayed Intervention group will serve as a control, receiving no intervention. After the initial 12 weeks, they will be entered into daily engagement with the HippoCamera app.
  Interventions: Behavioral: Memory replay

INTERVENTIONS:
Behavioral: Memory replay — Within the HippoCamera application, half of all recorded events will be categorized as "baseline" memories, and half will be categorized as "replay" memories.
  Baseline memories are recorded, but never viewed by the participant again until the "Early HippoCamera" test at the end of the 12-week intervention.
  Replay memories are recorded, and then placed into a memory gallery. HippoCamera uses a research-based algorithm to select 5 memories from this gallery for participants to replay each day. Prior research has shown that this replay is associated with significant memory enhancements for replayed v. baseline memories for HippoCamera users from other populations.

SUMMARY:
Down syndrome is a chromosomal abnormality associated with significant deficits across multiple cognitive domains, including a disproportionate deficit in hippocampally-dependent memory. In other words, individuals with Down syndrome may have a particular difficulty remembering specific details from past events. One way this manifests itself is in overgeneral autobiographical memory, or a tendency to remember the general gist of an event or cluster of events, rather than a single, isolated event. This overgeneral memory makes it difficult for individuals with Down syndrome to access their past, can interfere with attempts to becoming more independent, and increases anxiety and depression.

In the current VIRTUAL study, the investigators test whether a new digital memory prosthetic-HippoCamera-can enhance specific autobiographical memory in individuals with Down syndrome. In HippoCamera, users are asked to record and replay events from their daily lives. This replay is curated by a research-based algorithm in HippoCamera that optimizes consolidation of these events over time and has been shown to enhance memory specificity in other populations with memory impairments, particularly those that stem from hippocampal disfunction. It is, therefore, likely that similar enhancements in autobiographical memory specificity will be identified in individuals with Down syndrome, highlighting the benefits of this applications in this population.

DETAILED DESCRIPTION:
Individuals with Down syndrome exhibit a disproportionate deficit in hippocampally-dependent memory, including a particular difficulty remembering event-specific details of events from their own lives (i.e., autobiographical memory). In the proposed research, the investigators test the efficacy of a digital memory prosthetic-the HippoCamera application-in supporting this specific autobiographical memory in individuals with Down syndrome. In HippoCamera, participants are asked to record one event each day and replay up to five recorded events from prior days. This replay is curated by a research-based algorithm in HippoCamera that optimizes consolidation of these events over time. HippoCamera replay has been shown to enhance memory specificity in other populations with memory impairments, particularly those that stem from hippocampal disfunction. Specifically, memories that were replayed during the intervention were remembered with greater specificity than those that were just recorded and not replayed. The current research attempts to extend these findings by showing memory enhancements in a population with intellectual disabilities. Specifically, there are two independent aims:

Goal 1: Does using HippoCamera to record and replay daily events lead to greater memory specificity for the replayed events? To test the efficacy of HippoCamera in enhancing replayed memories, the current study compares memory for replayed and not replayed events in a sample of 40 individuals with Down syndrome. All participants enrolled in the study will take part in this intervention, allowing a within-subject comparison of replayed vs. not replayed events. This difference will be tested at two points: immediately (right after the 12-week intervention) and delayed (6 weeks after the 12-week intervention).

Goal 2: Does using HippoCamera to record and replay daily events help participants to develop memory-oriented strategies and behaviors that lead to global memory improvements?

It is possible that the greater benefit of HippoCamera is a global memory enhancement for all autobiographical memories in individuals who complete the intervention. To explore global memory benefits, the 40 participants will be pseudo-randomly assigned to one of two intervention groups (20 each in Groups A and B; pseudo-randomized to ensure matching of age, education, and baseline memory performance).

Critically, although all participants will eventually take part in the intervention, Group B will have a delayed start. In other words, all participants will complete the baseline memory test at the time of enrollment, then participants in Group A will immediately begin the intervention while participants in Group B will serve as a no-intervention control. At the end of Group A's 12-week intervention, both groups will complete a follow-up memory test.

Baseline-to-follow-up increases in memory specificity in Group A (i.e., intervention arm) will be compared to the same increases in Group B (i.e., control arm); greater increases in Group A could then be attributed to their enrollment in the 12-week intervention).

After serving as the control group for Group A's 12-week intervention, Group B will then begin the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Down syndrome
* Daily access to a smart phone
* The ability to create and replay memories using HippoCamera with limited support from a guardian
* Informed consent obtained from parent or guardian (or participant, if legally independent)
* Informed verbal assent obtained from participant
* Ability to comprehend instructions, denoted by parent/guardian acknowledgment
* English as a primary written and spoken language
* Normal or corrected-to-normal vision and hearing
* All races/ethnicities and socio-economic statuses

Exclusion Criteria:

* Autism
* Non-native speaker of English (acquired after the age of 5)

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Internal detail | Baseline memory appointment (immediately prior to intervention), immediate post-treatment appointment (within a week of terminating intervention), and follow-up appointment (6 weeks after terminating intervention).
  All memory narratives will be transcribed and scored using the Autobiographical Interview protocol.
  Highly trained raters will score each autobiographical memory according to the number and proportion of episodic (internal) vs. semantic (external) details. Episodic details are specific to the time and place of the targeted event, whereas semantic details involve factual information or extended events that do not require recollection of a specific time and place. Memory for episodic details requires the hippocampus, whereas memory for semantic details is more resistant to hippocampal damage.

SECONDARY OUTCOMES:
Positive memory content | Baseline memory appointment (immediately prior to intervention), immediate post-treatment appointment (within a week of terminating intervention), and follow-up appointment (6 weeks after terminating intervention).
  All memory narratives will be transcribed and scored using a text-based sentiment analysis (Valence Aware Dictionary and sEntiment Reasoner; VADER). VADER uses natural language processing to generate a weighted composite score of each narrative's overall sentiment between -1 (highly negative) to +1 (highly positive).
Independence | Baseline memory appointment (immediately prior to intervention), immediate post-treatment appointment (within a week of terminating intervention), and follow-up appointment (6 weeks after terminating intervention).
  Researchers will ask guardians to complete a brief survey describing participant independence. This survey will include questions about activities outside the house (e.g., work or school), social networks, and ability to perform self-care activities (e.g., feeding, dressing, etc.) independently. This survey will have a range of 0-20, with 20 indicating greater independence
Positive and Negative mood | Baseline memory appointment (immediately prior to intervention), immediate post-treatment appointment (within a week of terminating intervention), and follow-up appointment (6 weeks after terminating intervention).
  Participants will complete the Positive and Negative Affective Schedule (PANAS), a measure of positive and negative affect that has previously been used to evaluate mood in intellectual disability. The PANAS is a 20-item self-report questionnaire with 10 positive affect feelings/emotions and 10 negative affect feelings/emotions with possible scores ranging from (lowest) 20 to (highest) 100.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston College ONLINE STUDY, Chestnut Hill, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
All data will be anonymized prior to sharing. De-identified data from surveys will consist of tab-delimited output from the programs running the tasks. These data will be exported to a format that can be shared with researchers with either Macintosh or Windows platforms (e.g., .xls or .txt format). These files are small and should easily be able to be shared electronically with interested researchers, via email or secure servers.
  Videos and transcribed narratives of memories will not be shared, but scored data (e.g., detail and positivity scores) for each memory will be easily de-identified and saved as an excel file on a secure server. These de-identified scored data files will be small and should easily be able to be shared electronically with interested researchers, via email or secure servers.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Deidentified data will be available for access and sharing with interested researchers as soon as the final version of the manuscript is accepted for publication.
Access Criteria: Survey data and autobiographical memory scores will be uploaded to a public database (e.g., OSF) in conjunction with each publication.